CLINICAL TRIAL: NCT04098159
Title: Role of Regular Surveillance on Maintenance of Patency of an Arteriovenous Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Rashed, resident of vascular surgery, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Surveillance of an A-V access
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Hemodialysis Access Failure
MeSH Terms: interventions — Ultrasonography, Doppler, Duplex; Angioplasty; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESRD Patients have functioning or failing VAs (AVFs or AVGs). (Experimental)
  Interventions: Device: duplex ultrasound

INTERVENTIONS:
Device: duplex ultrasound — regular duplex follow up every three months with subsequent intervention either diagnostic venography , angioplasty or surgery according to the type of the lesion
  Other Names: diagnostic venography; angioplasty; surgery

SUMMARY:
Chronic Kidney disease (CKD) is a worldwide public health problem that classified into five stages (1). End stage renal disease (CDK stage 5) patients require a well-functioning vascular access (VA) for successful hemodialysis treatment (2). Types of VA include arteriovenous fistulae (AVFs) and arteriovenous grafts (AVGs). A vascular access is liable to early or late complications, and ultimately access failure. A meta-analysis showed that a 17% mean early access failure However recent studies have shown higher failure rates of up to 46%, with one year patencies between 52% to 83% (3). Low VA flow, thrombosis and loss of patency may result in under-dialysis that leads to increased morbidity, mortality and healthcare expenditure (4). In the majority of VAs, stenoses develop over variable intervals causing VA thrombosis and failure (5). If early detected and corrected, VA function and patency can be preserved and under-dialysis can be minimized or avoided. The aim of this study is to find out the role of periodic surveillance of VA in the detection of VA dysfunction and correctable lesions that may necessitate pre-emptive interventions to maintain VA patency and prevent VA loss

ELIGIBILITY:
Inclusion Criteria:

* ESRD Patients have functioning or failing VAs (AVFs or AVGs).

Exclusion Criteria:

* ESRD patients have infected or failed VAs .
* patientrefusal .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Number, type and technical success rate for elective interventions | within one year of creation of the VA

SECONDARY OUTCOMES:
secondary patency rate of the Arteriovenous Access after elective intervention | within one year of creation of the VA
number , type of complication that resulted from elective interventions | within one year of creation of the VA
primary patency rate of newly created Arteriovenous Access in assiut governorate | within one year of creation of the VA

REFERENCES:
- [Background] Gray RJ, Sacks D, Martin LG, Trerotola SO. Reporting standards for percutaneous interventions in dialysis access. Technology Assessment Committee. J Vasc Interv Radiol. 1999 Nov-Dec;10(10):1405-15. doi: 10.1016/s1051-0443(99)70252-6. No abstract available. PMID 10584659
- [Background] Lee T, Mokrzycki M, Moist L, Maya I, Vazquez M, Lok CE; North American Vascular Access Consortium. Standardized definitions for hemodialysis vascular access. Semin Dial. 2011 Sep-Oct;24(5):515-24. doi: 10.1111/j.1525-139X.2011.00969.x. Epub 2011 Sep 9. PMID 21906166
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Hakim RM, Breyer J, Ismail N, Schulman G. Effects of dose of dialysis on morbidity and mortality. Am J Kidney Dis. 1994 May;23(5):661-9. doi: 10.1016/s0272-6386(12)70276-7. PMID 8172208
- [Background] Tordoir J, Canaud B, Haage P, Konner K, Basci A, Fouque D, Kooman J, Martin-Malo A, Pedrini L, Pizzarelli F, Tattersall J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG on Vascular Access. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii88-117. doi: 10.1093/ndt/gfm021. No abstract available. PMID 17507428
- [Background] Besarab A. Advances in end-stage renal diseases 2000. Access monitoring methods. Blood Purif. 2000;18(4):255-9. doi: 10.1159/000014445. No abstract available. PMID 10965064